CLINICAL TRIAL: NCT01577342
Title: Determining the Effect of Antibiotic Drop Prophylaxis on the Conjunctival Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Healthcare Foundation (Other)
Responsible Party: Principal Investigator, Phil Hooper, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-10-458; 17354 (Other: REB)
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin 0.5% (Active Comparator): 1 drop four times daily for 3 days in affected eye post intravitreal injection
  Interventions: Drug: Moxifloxacin 0.5%
- No antibiotic use (No Intervention)

INTERVENTIONS:
Drug: Moxifloxacin 0.5% — 1 drop 4 times daily times 3 days post ranibizumab intravitreal injection
  Other Names: Vigamox
  Arms: Moxifloxacin 0.5%

SUMMARY:
Ranibizumab (Lucentis) is currently the best treatment for wet Age-Related Macular Degeneration (AMD). To work, the drug must be injected by means of an intravitreal injection (IVT) into the vitreous (jelly-like material) cavity in the back of the eye, repeatedly at intervals ranging from one to several months. Endophthalmitis is a rare but devastating infection of the eye that occurs in approximately 0.2% of patients after IVT injection. Many ophthalmologists ask patients to use antibiotic eye drops after IVT injection in the hope that this may reduce the risk of endophthalmitis. There is no proof that this happens and there is a possible risk that repeated exposure to the same antibiotic may cause antibiotic resistance organisms (bacteria) to develop over time.

The investigators hypothesize that repeated exposure to antibiotic during the initial stages of treatment for AMD will result in a progressive shift in the conjunctival flora with an increasing number of antibiotic resistant organisms appearing over time. If this is demonstrated, changes to the prevailing treatment approach will be needed to reduce the long term risk of a patient developing antibiotic resistant endophthalmitis during treatment.

DETAILED DESCRIPTION:
Intraocular injection of a VEGF inhibitor on a repeated basis has become the standard of care for the treatment of Age-Related Macular Degeneration (AMD) following pivotal studies which demonstrated that vision could be stabilized in 90% of treated patients. Most patients require injection, on average, every two months indefinitely.

The incidence of intraocular infection (endophthalmitis) following intraocular injection is approximately 0.2%. Current injection protocols involve the use of topical poviodine prior to injection based on evidence that this significantly reduces the bacterial flora on the conjunctiva. Following injection there is often some reflux of vitreous fluid from the cavity of the eye into the subjunctival space. For this reason many Ophthalmologists have patients use topical antibiotics for 2-3 days post injection with the expectation that this may reduce the risk of infection as the eye is healing.

Ta et al have demonstrated that following a 3 day course of topical antibiotic the incidence of resistant strains of bacteria in the conjunctival sac does not significantly increase (159 patients).There are no longitudinal studies which examine the effects of repeated short term antibiotic exposure on the conjunctival flora over time.

This is a prospective, randomized, comparative study which will follow the conjunctival flora of patients undergoing induction treatment with a VEGF inhibitor for AMD. The incidence of resistant organisms in the group receiving antibiotics will be compared to that in a similar group who do not receive antibiotics. Following informed consent, patients will have a conjunctival swab taken by the treating Ophthalmologist after instillation of sterile topical anesthetic but before application of poviodine. The swabs will be cultured in thyoglycollate broth. Bacteria present and resistance to the antibiotic used will be identified. This process will be repeated each visit during the induction phase of treatment which consists of four sequential injections each a month apart.

Patients in the antibiotic arm will be asked to use topical Moxifloxacin drops 4 times a day for 3 days following injection. The control group will not receive antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing their first ever injection to treat AMD and who are expected to continue treatment in London for at least the next 3 injections are potentially eligible.
* able to provide Informed Consent.

Exclusion Criteria:

* current contact lens use.
* use of topical antibiotics in the study eye in the preceding 6 months.
* patients in whom eye surgery in the study eye is anticipated in the next 4 months.
* documented allergy to the drug or vehicle.
* patients with active ocular, periocular or systemic infection.
* immunosuppressed patients.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic resistant organisms | 4 months
  Conjunctival culture will be obtained in the designated "study" eye prior to the first intravitreal injection in de novo AMD patients and will be repeated prior to the next 3 injections.
  Susceptibility or resistance of the ocular surface flora to Moxifloxicin will be assessed by standard micro analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Hooper, MD, FRCSC, Principal Investigator — Ivey Eye Institute, St. Joseph's Health Care Centre
Locations (1):
- Ivey Eye Institute, St. Joseph's Health Care Centre, London, Ontario, Canada